CLINICAL TRIAL: NCT02303730
Title: Exenatide BID Compared With Insulin Glargine to Change Liver Fat Content in Non-alcoholic Fatty-liver Disease Patients With Type 2 Diabetes
Brief Title: Exenatide Compared With Insulin Glargine to Change Liver Fat Content in Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: Huadong Hospital (Other); Shanghai Minhang Central Hospital (Other); Shanghai 6th People's Hospital (Other); Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Xin Gao, vice-president, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESR-14-10096
Record Dates: First submitted 2014-11-23; First posted 2014-12-01 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Diabetes Mellitus, Type 2; Non-alcoholic Fatty Liver Disease
Keywords: Diabetes; Non-alcoholic Fatty Liver Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Non-alcoholic Fatty Liver Disease; Diabetes Mellitus | interventions — Exenatide; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exenatide (Experimental): Exenatide 5 ug twice daily 1 hour before meal subcutaneously for 4 weeks, then add to 10 ug twice daily 1 hour before meal subcutaneously for another 20 weeks
  Interventions: Drug: Exenatide
- Insulin glargine (Active Comparator): Insulin glargine subcutaneously, once daily, for 24 weeks
  Interventions: Drug: insulin glargine

INTERVENTIONS:
Drug: Exenatide — The starting dose of exenatide is 5 ug bid, subcutaneously, for 4 weeks, followed by 10 ug bid, subcutaneously, for 20 weeks. If hypoglycaemia (blood glucose<2.9 mmol/l or < 3.9 mmol/l at least 2 times) or serious intolerance occurs, the dose will be adjusted to 5 ug bid, subcutaneously.
  Other Names: Byetta
  Arms: Exenatide
Drug: insulin glargine — The starting dose of insulin glargine will depend upon the HbA1c level at screening(HbA1c <8% use 0.1 -0.2 U/kg per day;HbA1c >8% use 0.2 -0.3 U/kg per day).
  Dose adjustment protocol for insulin glargine (at least 3 determinations of fasting blood glucose per week):
  fasting blood glucose(FBG) > 180 mg/dL(10 mmol/l): add 4 U; FBG 140-180 mg/dL(7.8-10 mmol/l): add 2 U; FBG 126-139 mg/dL(7.0-7.8 mmol/l): add 1 U.
  If hypoglycemia, reduce insulin glargine by:
  blood glucose <70mg/dl（3.9mmol/l）: 10%-20%; blood glucose <40mg/dl（2.2mmol/l）: 20%-40%.
  Other Names: Lantus
  Arms: Insulin glargine

SUMMARY:
The purpose of this study is to evaluate whether exenatide is superior to insulin glargine (after 24 weeks) in reducing liver fat content (by MRS) in patients with newly diagnosed type 2 diabetes mellitus and concomitant non-alcoholic fatty-liver disease(NAFLD).

DETAILED DESCRIPTION:
This is a randomized, open-label, parallel-group, active controlled, multi-center clinical trial to investigate whether exenatide is superior to insulin glargine in reducing liver fat content in patients with newly diagnosed type 2 diabetes mellitus and concomitant NAFLD.Patients with type 2 diabetes and concomitant NAFLD from 18-70 years of age, with inadequate glycaemic control defined as 7% ≤ HbA1c ≤ 10% and BMI≥24kg/ m2 at the time of screening. Patients should be on diet and exercise but drug treatment naive, no use of any glucagon-like peptide-1(GLP-1) analogues or insulin within 3 months before enrolment.Patients will have an screening period 2 weeks, and a 24-week open label treatment period.

All demographic data variables collected by descriptive analysis tests are used. Qualitative variables use absolute frequency and percentage, and numeric variables use average, mean, median, standard deviation, maximum, minimum, quartiles, etc. Unless specifically stated, statistical significance will be defined as P<0.05 in the whole analysis procedure.For the primary endpoint of this study, superiority test will be applied to the quantitative data of these two groups. For secondary and exploratory efficacy variables, difference test will be used to analyse repeated measurement data from two groups. For essential Safety parameters, difference test will be used to analyse the differences between two groups.The analysis of all primary and secondary endpoints of efficacy and safety must be based on the Full Analysis Set (FAS). As supporting evidence, the analysis of primary endpoint variables must also comply with the Pre-protocol (PPS) Analysis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 ≤ age ≤ 70 years old.
* Newly diagnosed type 2 diabetes mellitus (WHO Diagnostic criteria for diabetes mellitus, 1999).
* Patients with NAFLD, MRS measurement of liver fat content> 10%.
* 7% ≤ HbA1c ≤ 10%
* No heavy drinking history within the last 5 years (alcohol intake: male < 20 g/d, female < 10 g/d)
* HBsAg (-), hepatitis C virus antibody (HCV-Ab) (-)
* BMI ≥ 24 kg/m2;

Exclusion Criteria:

* Pregnancy, lactation, intended pregnancy, or failure to take adequate contraceptive measures taken (contraception measures including sterilization, intrauterine device, oral contraceptives, and persistent use of condoms).
* Type 1 diabetes mellitus, gestational diabetes mellitus or other special types of diabetes.
* Liver and renal dysfunction (ALT or aspartate aminotransferase(AST) is 2.5 times higher than the upper limit of normal, or total bilirubin is 1.5 times higher than the upper limit of normal, or Cr ≥ 115 μmol/L).
* increased amylase (blood amylase is 2.5 times higher than the upper limit of normal) or presence of gastrointestinal disease.
* Use of drugs that may affect liver fat content within one month before or during the trial period, such as glucocorticoids, thyroid hormone, etc.
* Use of GLP-1 receptor agonist, dipeptidyl peptidase -4 (DPP-4) inhibitors or insulin within 3 months before enrolment
* Presence of serious dyslipidemia or other endocrine diseases (hypothyroidism, hypothalamic-pituitary dysfunction, etc).
* Fatty liver caused by viral hepatitis, drug, alcohol, Wilson disease or total parenteral nutrition.
* Presence of liver cancer, infection, biliary tract disease or recently increased liver enzyme due to medication.
* Participation in strenuous exercise or administration of any drugs that affect glucose metabolism.
* History of pancreatitis, alcohol abuse, metal disorders or history of allergy to investigational drug.
* Congestive heart failure defined as New York Heart Association (NYHA) class III or IV, unstable angina or myocardial infarction in recent 6 months.
* Any situation that may affect the implementation or results of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2015-03; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Change in liver fat content（%） measured by MRS | baseline and 24 weeks
  Change in liver fat content（%） measured by MRS

SECONDARY OUTCOMES:
Change in intra-abdominal visceral fat content (cm2), abdominal subcutaneous fat content (cm2), and ratio between intra-abdominal visceral fat and subcutaneous fat area by MRI | baseline and 24 weeks
  Change in intra-abdominal visceral fat content (cm2), abdominal subcutaneous fat content (cm2), and ratio between intra-abdominal visceral fat and subcutaneous fat area by MRI
Change in glucose metabolism (fasting blood glucose, postprandial plasma glucose, HbA1c) | baseline and 24 weeks
  Change in glucose metabolism (fasting blood glucose, postprandial plasma glucose, HbA1c)
Change in blood lipid profile (total cholesterol, triglyceride, HDL, LDL) | baseline and 24 weeks
  Change in blood lipid profile (total cholesterol, triglyceride, HDL, LDL)
Change in body weight,waist circumference and hip circumference | baseline and 24 weeks
  Change in body weight,waist circumference and hip circumference

OTHER OUTCOMES:
Change in cardiac function measured by echocardiography | baseline and 24 weeks
  Change in cardiac function measured by echocardiography
Change in β-cell function (fasting C-peptide, 2-hour postprandial C-peptide) | baseline and 24 weeks
  Change in β-cell function (fasting C-peptide, 2-hour postprandial C-peptide)
Change in liver enzymes and laboratory parameters (hematology, biochemical tests) | baseline and 24 weeks
  Change in liver enzymes and laboratory parameters (hematology, biochemical tests)
Incidence of hypoglycaemia events | up to 24 weeks
  Incidence of hypoglycaemia events
Incidence of adverse events（AEs）and Severe adverse events(SAEs) | up to 24 weeks
  Incidence of adverse events（AEs）and Severe adverse events(SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Xin Gao, doctor, Principal Investigator — Fudan University
Locations (5):
- China (5):
  - Department of Endocrinology and Metabolism, Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Department of Endocrinology and Metabolism, Shanghai Minhang Central Hospital, Shanghai, Shanghai Municipality
  - Department of Endocrinology and Metabolism,Huadong Hospital, Shanghai, Shanghai Municipality
  - Department of Endocrinology and Metabolism,Shanghai 6th People's Hospital, Shanghai, Shanghai Municipality
  - Department of Endocrinology and Metabolism,Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xu W, Bi Y, Sun Z, Li J, Guo L, Yang T, Wu G, Shi L, Feng Z, Qiu L, Li Q, Guo X, Luo Z, Lu J, Shan Z, Yang W, Ji Q, Yan L, Li H, Yu X, Li S, Zhou Z, Lv X, Liang Z, Lin S, Zeng L, Yan J, Ji L, Weng J. Comparison of the effects on glycaemic control and beta-cell function in newly diagnosed type 2 diabetes patients of treatment with exenatide, insulin or pioglitazone: a multicentre randomized parallel-group trial (the CONFIDENCE study). J Intern Med. 2015 Jan;277(1):137-50. doi: 10.1111/joim.12293. Epub 2014 Aug 5. PMID 25039675
- [Background] Gupta NA, Mells J, Dunham RM, Grakoui A, Handy J, Saxena NK, Anania FA. Glucagon-like peptide-1 receptor is present on human hepatocytes and has a direct role in decreasing hepatic steatosis in vitro by modulating elements of the insulin signaling pathway. Hepatology. 2010 May;51(5):1584-92. doi: 10.1002/hep.23569. PMID 20225248
- [Background] Sharma S, Mells JE, Fu PP, Saxena NK, Anania FA. GLP-1 analogs reduce hepatocyte steatosis and improve survival by enhancing the unfolded protein response and promoting macroautophagy. PLoS One. 2011;6(9):e25269. doi: 10.1371/journal.pone.0025269. Epub 2011 Sep 21. PMID 21957486
- [Background] Okerson T, Yan P, Stonehouse A, Brodows R. Effects of exenatide on systolic blood pressure in subjects with type 2 diabetes. Am J Hypertens. 2010 Mar;23(3):334-9. doi: 10.1038/ajh.2009.245. Epub 2009 Dec 17. PMID 20019672
- [Background] Cuthbertson DJ, Irwin A, Gardner CJ, Daousi C, Purewal T, Furlong N, Goenka N, Thomas EL, Adams VL, Pushpakom SP, Pirmohamed M, Kemp GJ. Improved glycaemia correlates with liver fat reduction in obese, type 2 diabetes, patients given glucagon-like peptide-1 (GLP-1) receptor agonists. PLoS One. 2012;7(12):e50117. doi: 10.1371/journal.pone.0050117. Epub 2012 Dec 6. PMID 23236362
- [Background] Kenny PR, Brady DE, Torres DM, Ragozzino L, Chalasani N, Harrison SA. Exenatide in the treatment of diabetic patients with non-alcoholic steatohepatitis: a case series. Am J Gastroenterol. 2010 Dec;105(12):2707-9. doi: 10.1038/ajg.2010.363. No abstract available. PMID 21131943
- [Background] Sathyanarayana P, Jogi M, Muthupillai R, Krishnamurthy R, Samson SL, Bajaj M. Effects of combined exenatide and pioglitazone therapy on hepatic fat content in type 2 diabetes. Obesity (Silver Spring). 2011 Dec;19(12):2310-5. doi: 10.1038/oby.2011.152. Epub 2011 Jun 9. PMID 21660077
- [Background] Shao N, Kuang HY, Hao M, Gao XY, Lin WJ, Zou W. Benefits of exenatide on obesity and non-alcoholic fatty liver disease with elevated liver enzymes in patients with type 2 diabetes. Diabetes Metab Res Rev. 2014 Sep;30(6):521-9. doi: 10.1002/dmrr.2561. PMID 24823873
- [Background] Juurinen L, Tiikkainen M, Hakkinen AM, Hakkarainen A, Yki-Jarvinen H. Effects of insulin therapy on liver fat content and hepatic insulin sensitivity in patients with type 2 diabetes. Am J Physiol Endocrinol Metab. 2007 Mar;292(3):E829-35. doi: 10.1152/ajpendo.00133.2006. Epub 2006 Nov 7. PMID 17090752
- [Background] ORIGIN Trial Investigators; Gerstein HC, Bosch J, Dagenais GR, Diaz R, Jung H, Maggioni AP, Pogue J, Probstfield J, Ramachandran A, Riddle MC, Ryden LE, Yusuf S. Basal insulin and cardiovascular and other outcomes in dysglycemia. N Engl J Med. 2012 Jul 26;367(4):319-28. doi: 10.1056/NEJMoa1203858. Epub 2012 Jun 11. PMID 22686416
- [Derived] Liu L, Wang R, Gao J, Yan J, Zhang J, Zhang Z, Liu J, Lin H, Rao S, Yao X, Wu W, Bian H, Wang X, Guo S, Gao X, Yan H. Insulin Glargine is More Suitable Than Exenatide in Preventing Muscle Loss in Non-Obese Type 2 Diabetic Patients with NAFLD. Exp Clin Endocrinol Diabetes. 2023 Nov;131(11):583-588. doi: 10.1055/a-2145-1004. Epub 2023 Jul 31. PMID 37524110